CLINICAL TRIAL: NCT01906112
Title: Role of Surgery for the Primary in Patients With Breast Cancer Stage IV - A Prospective Randomized Multicenter Controlled Trial
Brief Title: Role of Surgery for the Primary in Patients With Breast Cancer Stage IV.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual and no further funding.
Sponsor: National Cancer Institute, Thailand (Other Government)
Collaborators: Vichaiyut Hospital (Other)
Responsible Party: Principal Investigator, AKANIST PIYAPANT, MD.,FRCST., Surgical Oncologist., National Cancer Institute, Thailand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17_2013RC_IN305
Record Dates: First submitted 2013-07-15; First posted 2013-07-23 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Carcinoma Breast Stage IV
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Controlled (No Intervention): No surgery for primary breast tumor.
- Study (Experimental): Surgery for primary breast tumor.
  Interventions: Procedure: Surgery for primary breast tumor.

INTERVENTIONS:
Procedure: Surgery for primary breast tumor. — Complete resection of primary breast tumor(Lumpectomy or mastectomy)
  Arms: Study

SUMMARY:
The purpose of this study is to determine benefits of surgery for the primary in patients with breast cancer stage IV in randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy breast cancer stage IV patients with resectable primary breast tumor.
* Resectable breast cancer stage IV patients who well response of visceral metastasis to systemic therapy and fit for surgery.

Exclusion Criteria:

* Breast cancer stage IV patients with local complication of primary breast tumor that require surgery for palliation such as uncontrolled bleeding,large and non-healing ulcer or intractable pain.
* Breast cancer stage IV patients with unresectable primary breast tumor or extensive chest wall disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Five years

SECONDARY OUTCOMES:
Quality of life & Uncontrolled chest wall disease | Five years

CONTACTS AND LOCATIONS:
Overall Officials: AKANIST PIYAPANT, MD.,FRCST., Principal Investigator — Phyathai2 Hospital , Bangkok, Thailand
Locations (9):
- Thailand (9):
  - Division Head & Neck and Breast, Department of Surgery. Faculty of Medicine Siriraj Hospital, Bangkok Noi, Bangkok
  - Department of Surgery, Faculty of Medicine Vajira Hospital., Dusit, Bangkok
  - Phyathai 2 Hospital, PhyaThai, Bangkok
  - National Cancer Institute, Ratchathewi, Bangkok
  - Phramongkutklao Hospital, Ratchathewi, Bangkok
  - Chonburi Cancer Hospital, Muang Chonburi, Changwat Chon Buri
  - Khon Kaen University, Muang, Changwat Khon Kaen
  - Suratthani Cancer Hospital, Muang Suratthani, Changwat Surat Thani
  - Udon Thani Cancer Hospital, Muang Udon Thani, Changwat Udon Thani

REFERENCES:
- [Background] Khan SA, Stewart AK, Morrow M. Does aggressive local therapy improve survival in metastatic breast cancer? Surgery. 2002 Oct;132(4):620-6; discussion 626-7. doi: 10.1067/msy.2002.127544. PMID 12407345
- [Background] Gnerlich J, Jeffe DB, Deshpande AD, Beers C, Zander C, Margenthaler JA. Surgical removal of the primary tumor increases overall survival in patients with metastatic breast cancer: analysis of the 1988-2003 SEER data. Ann Surg Oncol. 2007 Aug;14(8):2187-94. doi: 10.1245/s10434-007-9438-0. Epub 2007 May 24. PMID 17522944
- [Background] Rapiti E, Verkooijen HM, Vlastos G, Fioretta G, Neyroud-Caspar I, Sappino AP, Chappuis PO, Bouchardy C. Complete excision of primary breast tumor improves survival of patients with metastatic breast cancer at diagnosis. J Clin Oncol. 2006 Jun 20;24(18):2743-9. doi: 10.1200/JCO.2005.04.2226. Epub 2006 May 15. PMID 16702580
- [Background] Shien T, Kinoshita T, Shimizu C, Hojo T, Taira N, Doihara H, Akashi-Tanaka S. Primary tumor resection improves the survival of younger patients with metastatic breast cancer. Oncol Rep. 2009 Mar;21(3):827-32. PMID 19212646
- [Background] Neuman HB, Morrogh M, Gonen M, Van Zee KJ, Morrow M, King TA. Stage IV breast cancer in the era of targeted therapy: does surgery of the primary tumor matter? Cancer. 2010 Mar 1;116(5):1226-33. doi: 10.1002/cncr.24873. PMID 20101736
- [Background] Nguyen DH, Truong PT, Alexander C, Walter CV, Hayashi E, Christie J, Lesperance M. Can locoregional treatment of the primary tumor improve outcomes for women with stage IV breast cancer at diagnosis? Int J Radiat Oncol Biol Phys. 2012 Sep 1;84(1):39-45. doi: 10.1016/j.ijrobp.2011.11.046. Epub 2012 Feb 11. PMID 22330986